CLINICAL TRIAL: NCT02880943
Title: Phase I/II Dose-finding, Safety and Efficacy Study of Radium-223 Dichloride (XOFIGO®) in Renal Cell Carcinoma Patients With Bone Metastases.
Brief Title: Dose-finding, Safety and Efficacy Study of Radium-223 Dichloride (XOFIGO) in RCC Patients With Bone Metastases. (EIFFEL)
Acronym: EIFFEL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Association Pour La Recherche des Thérapeutiques Innovantes en Cancérologie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EIFFEL
Record Dates: First submitted 2016-08-18; First posted 2016-08-26 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Clear-cell Metastatic Renal Cell Carcinoma; Bone Metastases
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma | interventions — radium Ra 223 dichloride; Radium-223

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Group A: patients with bone disease mainly will be treated with XOFIGO® alone.
  Node and/or adrenal metastases and/or ≤5 lung metastases ≤1cm each are allowed in Group A.
  Interventions: Drug: XOFIGO
- Group B (Experimental): Group B: patients already treated with an ongoing approved Tyrosine Kinase Inhibitor (TKI) for their visceral metastases will be treated with XOFIGO® for bone disease.
  Interventions: Drug: XOFIGO

INTERVENTIONS:
Drug: XOFIGO — XOFIGO® will be administered intravenously as a bolus injection every 4 weeks with a maximum of 6 administrations per patient.
  Four dose levels are available for evaluation : 27.5 kBq/kg, 55 kBq/kg, 88 kBq/kg and 110 kBq/kg.
  Starting dose for phase I will be 55 kBq/kg.
  Other Names: radium-223

SUMMARY:
This is a prospective, multicentre, open-label, phase I/II study to evaluate the maximum tolerated dose (MTD), and the most successful dose (MSD) of XOFIGO®, in renal cancer patients with metastases to bone, without (Group A) or with (Group B) visceral metastases.

DETAILED DESCRIPTION:
This is a prospective, multicentre, open-label, phase I/II study to evaluate the maximum tolerated dose (MTD), and the most successful dose (MSD) of XOFIGO®, in renal cancer patients with metastases to bone, without (Group A) or with (Group B) visceral metastases.

Dose-finding will be performed according to the Continual Reassessment Method (CRM) using either toxicity (escalation cohort) or joined toxicity-efficacy (expansion cohort) endpoints.

Two groups of patients will be evaluated:

* Group A: patients with bone disease mainly will be treated with XOFIGO® alone. (node and/or adrenal metastases and/or ≤5 lung metastases ≤1cm each are allowed in Group A).
* Group B: patients already treated with an ongoing approved Tyrosine Kinase Inhibitor (TKI) for their visceral metastases will be treated with XOFIGO® for bone disease.

XOFIGO® will be administered intravenously as a bolus injection every 4 weeks with a maximum of 6 administrations per patient. Four dose levels are available for evaluation : 27.5 kBq/kg, 55 kBq/kg, 88 kBq/kg and 110 kBq/kg.

Starting dose for phase I will be 55 kBq/kg.

Visit schedule:

Selection Patients will come to the hospital at baseline, and screening assessments must be performed within 28 days prior to first XOFIGO® administration.

XOFIGO® period Patients will receive an injection of XOFIGO® on Day 1 of each 4 weeks-cycle for a maximum of 6 cycles. Patients will be subject to physical examination, blood sampling and pain evaluation prior to each injection. Scintigraphy of biodistribution of radium-223 dichloride will be realised on C1D1 after the 1st injection of XOFIGO® On C1D15, patients will also come for physical examination and blood sampling. On C2D15 (end of DLT period for phase I), patients will also come for end of DLT period evaluation and will be subject to physical examination and blood sampling.

Prior to C3D1 and C5D1, patients will undergo WB-IRM and FNa-PET. End of treatment visit (EOT) will take place 4 weeks after the last administration of XOFIGO®.

In the absence of confirmed bone progression at XOFIGO® discontinuation time, patients will continue to undergo WB-IRM and FNa-PET every 2 months until confirmed bone progression or end of follow-up.

Confirmation of bone progression upon WB-IRM will be performed 4 weeks after the initial progression is observed.

Follow-up Patients will be followed-up for a maximum of 12 months from the 1st administration of XOFIGO®.

Number of subjects:

Maximum number of patients to be enrolled in the escalation cohort is 21. Maximum number of patients to be enrolled in the expansion cohort is 21. Group A: 2-4 patients; Group B: 38-40 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic renal cell carcinoma with a clear cell component.
2. Bone metastases upon bone scan with no CT and MRI performed any time within period of 4 weeks prior to study entry, with at least one evaluable unidimensional bone lesion (i.e., ≥1 malignant tumour mass that can be accurately measured in at least 1 dimension ≥ 10 mm on T1-weighted Magnetic Resonance Imaging [MRI]).

   Group A: bone metastases (lymph nodes and/or adrenal metastases, and/or ≤ 5 lung metastases of less than 1 cm each, are allowed).

   Group B: bone metastases AND visceral metastases upon MRI (according to revised RECIST 1.1 criteria).
3. Patient in a) first (naïve), or b) second or third line setting receiving or about to receive an approved Tyrosine Kinase Inhibitor (patients on mTOR inhibitors are not eligible).
4. Male or female, age ≥18 years at ICF signature time.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Good or Intermediate prognostic group according to the International Metastatic Database Consortium (IMDC).
7. At least 4 weeks from the end of a previous systemic treatment, if any, with resolution of all treatment-related toxicity according to NCI CTCAE Version 4.03 grade ≤ 1 except for alopecia.
8. Palliative local treatment allowed if performed ≥ 2 weeks prior to study entry for radiotherapy, cementoplasty or minor surgery; ≥ 4 weeks prior to study entry for major surgery.
9. Adequate organ function defined by the following criteria:

   * Absolute Neutrophils count (ANC) ≥1 500 cells/mm3
   * Platelets ≥100 000 cells/mm3
   * Haemoglobin ≥ 9.0 g/dL
   * AST and ALT ≤ 2.5 x upper limit of normal (ULN), unless there are liver metastases in which case AST and ALT ≤5.0 x ULN
   * Total bilirubin ≤ 1.5 x ULN
   * Estimated glomerular filtration rate upon MDRD ≥ 50 mL/min
   * Urinary protein < 2+ by urine dipstick. If dipstick is ≥ 2+ then a 24-hour urine collection can be done and the patient may enter only if urinary protein is < 2 g per 24 hours
   * Corrected calcium ≤ 2.8 mmol/L.
10. Women of childbearing potential must have a negative serum pregnancy test within 7days prior to treatment initiation.
11. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrolment.
12. Willingness, for men and women,to use effective contraception during study treatment and for 6 months after last dose of study drug.
13. Willingness to comply with protocol requirements.

Exclusion Criteria:

Poor prognostic group according to the IMDC. 2. Prior radiotherapy to ≥ 40% of bone marrow, whole pelvic irradiation and/or prior isotope therapy whatever the isotope (any α- or β-emitters).

3. Active secondary cancer including prior malignancy from which the subject has been disease-free for ≤ 3 years (however, adequately treated superficial basal cell skin or cervical carcinoma in situ before 4 weeks prior to entry are eligible to the study).

4. Known brain or leptomeningeal involvement. 5. Any other concurrent serious illness or medical conditions including:

* Crohn"s disease or ulcerative colitis
* Bone marrow dysplasia
* Known presence of osteonecrosis of the jaw 6. Uncontrolled hypertension. 7. Uncontrolled cardiac arrhythmias, angina pectoris, and/or hypertension. History of congestive heart failure, or myocardial infarction within the last 6 months.

  8. QTc interval (QTc) assessed by local device > 500ms in the 7 days prior to inclusion.

  9. Ongoing biphosphonates, denosumab and/or vitamin D supplementation. 10. Active infection requiring systemic antibiotic or anti-fungal medication. 11. Any contra-indication to MRI, including:
* Carrying a metallic medical device (e.g. pacemaker) or foreign body prohibiting use of MRI
* Known allergy to gadolinium or iodine
* Dysthyroidism precluding usage of iodine contrast agent 12. Pregnant or breast feeding. 13. Participation in another clinical trial with any investigational drug within 30 days prior to study enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2016-10; Primary Completion 2020-10 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLT) | within 6 weeks after the first injection of XOFIGO
  Dose-limiting toxicities (DLT) within the first 6 weeks to determine the MTD.
  DLT is defined as any XOFIGO related adverse event occurring between C1D1 and C2D15.

SECONDARY OUTCOMES:
Distribution of radium-223 dichloride into the bone assessed with scintigraphy of biodistribution of radium-223 dichloride | Assessed at day 1 after the first Xofigo injection
  Distribution of radium-223 dichloride into the bone assessed with scintigraphy of biodistribution of radium-223 dichloride
Bone response concordance between FNa-PET scan and whole-body MRI | up to 12 months
Bone clinical benefit rate (bone objective response or stable disease, BCB) | up to 12 months
Overall clinical benefit rate (bone and visceral objective response or stable disease, OCB) | up to 12 months
Changes in bone markers | up to 12 months
  Changes in bone markers: bone formation: bone alkaline phosphatase [bALP], N-terminal type I collagen [PINP]; bone resorption: C-terminal telopeptide cross-linking of type I collagen [S-CTX-I], cross-linked C-terminal telopeptide of type I collagen [ICTP]), TRACP 5b, sRANKL, osteoprotegerin (OPG)
Time to occurrence of the first Skeletal-Related Events (SRE) | up to 12 months
  SRE including pathological fracture, requirement to initiate radiotherapy, spinal cord compression or requirement for bone surgery
Time to bone progression (TTBP) defined as the time from the first administration of XOFIGO® to the bone tumour progression (revised RECIST 1.1 taking into account bone lesions) | up to 12 months
1-year overall survival rate (1y-OS) defined as the percentage of patients alive 1 year after 1st administration of XOFIGO® | 1 year
Pain assessment upon Brief Pain Inventory (BPI) and analgesic consumption questionnaire | BPI questionnaire will be completed 7 days before the first administration of XOFIGO® and before each visit.
Change From Baseline in the FACT-Kidney Symptom Index-15 (FKSI-15) Scale | 7 months (Baseline and at 7 months)
  FKSI-15 questionnaire will be performed only for patients included in the phase II part of the study.
Changes in MRI | up to 12 months
  New MRI criteria as prediction markers for progression and for disease specific and overall survival:
  Diffusion weighted imaging (DWI): Apparent diffusion coefficient (ADC) values in the five target bone lesions
  * Ultra-short echo time (UTE) sequence: T2 measurements in the five target bone lesions
  * Perfusion weighted imaging (PWI): assessments of the area under the curve at 1min30, and of the focal lesion (FLE max) enhancement.
Change From Baseline in EQ-5D Scale | 7 months (Baseline and at 7 months)
  EQ-5D questionnaire will be performed only for patients included in the phase II part of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Stephane OUDARD, MD, Principal Investigator — Hôpital Européen Georges Pompidou, Oncology Department
Locations (5):
- France (5):
  - CHU Bordeaux (St. André), Bordeaux
  - Centre François Baclesse, Caen
  - Hôpital Cochin, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No